CLINICAL TRIAL: NCT00540709
Title: PUMP STUDY MDI Lantus/Lispro vs Continuous Insulin+Lispro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901 4036
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine

SUMMARY:
Whether a once-daily basal injection of insulin glargine with mealtime injections of insulin lispro achieves equivalent glycaemic control (HbA1c) to administration of insulin lispro by continuous subcutaneous insulin infusion in Type 1 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes mellitus for at least one year.
* Subjects with no previous experience with Continuous Subcutaneous Insulin Infusion (CSII) or insulin glargine,
* capable of managing a basal-bolus regimen and meeting glycaemic targets in accordance with the protocol.
* HbA1c > than or = to 6.5 < than or = to 9.0% at screening visit with evidence of lack of insulin secretion (e.g. fasting C-peptide concentration is < 0.1 nmol/l with fasting blood glucose(FBG) > 126 mg/dl).

Exclusion Criteria:

* Previous therapy using insulin glargine or continuous subcutaneous insulin infusion.
* Lipodystrophy preventing adequate use of CSII.
* Unwilling or unlikely to be able to use MiniMedr insulin pump with insulin lispro for CSII.
* Unwilling or unlikely to be able to use an MDI regimen with insulin glargine and insulin lispro in accordance with the protocol (for instance, subjects who routinely use a twice-daily mixed insulin regimen should not be included).
* History of more than two severe hypoglycaemic episodes in the past 6 months.
* Acute infection which, in the opinion of the investigator, could lead to increased insulin resistance.
* Acute or chronic metabolic acidosis.
* Episode of DKA (diabetic ketoacidosis) within the last three months.
* Active, uncontrolled, advanced diabetic retinopathy.
* Impaired hepatic function, as shown by > 2.5 times the upper limit of normal range for AST.
* Impaired renal function, as shown by serum creatinine > 1.5mg/dl.
* History of gastroparesis. Congestive heart failure requiring ongoing pharmacological treatment.
* Stroke, myocardial infarction (MI), coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) or angina pectoris within the last 12 months.
* Treatment with a non-selective beta blocker.
* Treatment with inhaled or systemic steroids.
* History of hypersensitivity to insulin lispro or to any drug with a similar chemical structure to insulin glargine or insulin lispro or to any of the excipients of the insulin glargine and insulin lispro preparations used in the study.
* Any malignancy within the last five years, except adequately treated basal cell carcinoma.
* History within the last two years or current addiction to substances of abuse including ethanol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2002-11; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Primary efficacy data was HbA1c. | At week 24 (the last day of the treatment period).

SECONDARY OUTCOMES:
Secondary efficacy data included HbA1c. | At Week 8 and Week 16 after starting study medication and selfmonitored blood glucose (SMBG) measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

REFERENCES:
- [Derived] Bolli GB, Kerr D, Thomas R, Torlone E, Sola-Gazagnes A, Vitacolonna E, Selam JL, Home PD. Comparison of a multiple daily insulin injection regimen (basal once-daily glargine plus mealtime lispro) and continuous subcutaneous insulin infusion (lispro) in type 1 diabetes: a randomized open parallel multicenter study. Diabetes Care. 2009 Jul;32(7):1170-6. doi: 10.2337/dc08-1874. Epub 2009 Apr 23. PMID 19389820